CLINICAL TRIAL: NCT03763474
Title: The Effect of Mobile Application Euglyca in Glycemic Control of Children and Adolescents With Diabetes Mellitus Type-1
Brief Title: Euglyca Application in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Christos Chatzakis, Christos Chatzakis MD, MSc, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Euglyca application
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors were blinded as for the allocation of the patients in the 2 groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Euglyca (Experimental): Patients randomized to the Euglyca group were advised to download the Euglyca application on their smartphones and they were asked to use the application for the calculation of the bolus insulin dose.
  Interventions: Combination Product: Euglyca application
- Control (No Intervention)

INTERVENTIONS:
Combination Product: Euglyca application — 'Euglyca' is a mobile application developed by two of the authors (CC and DF). The application has a data base of 7000 foods and food products met in greek eating habits as well as the corresponding amount of carbohydrates and lipids for each of them. Subsequently, the amount of carbohydrates and lipids contained in a meal are calculated automatically by the application. By taking into consideration the amount of carbohydrates and lipids to be consumed, the preprandial and target post-prandial glycemia concentrations, the insulin correction factor for the patient, the carbohydrates and lipids factors and the active insulin (in case of CSII), 'Euglyca' calculates the required bolus dose of insulin.
  Arms: Euglyca

SUMMARY:
80 children and adolescents with Diabetes Mellitus Type 1 were enrolled in the study and were randomly assigned in the intervention group (Euglyca group) or in the control group. Patients in the Euglyca group were asked to use the application in order to calculate the bolus insulin dose. Primary outcomes of the study were the Glycosylated hemoglobin, percentage of normoglycemias and the Diabetes Treatment Satisfaction Questionnaire Score. Patients were evaluated at the baseline, 3, 6 and 12 months after the beginning of the study.

DETAILED DESCRIPTION:
Children and adolescents with Diabetes Mellitus Type 1 (T1DM) who visited consecutively this clinic were asked to participate in the study if they owned an Android smartphone and were familiar with its use. Patients were included after one of their parents or their legal guardian signed an informed consent. Inclusion criteria were: 1. Treatment with multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII); 2. satisfactory knowledge of the concept of carbohydrates and lipids counting acquired following previous training by the physicians and nutritionist of the department at initial diagnosis and thereafter during follow-up visits. Exclusion criteria were: 1. Use of another medical application for diabetes in the previous 3 months; 2. lack of capacity of reading greek.

80 patients met the inclusion criteria and agreed to participate in the study. Subsequently they were randomized to two equally numbered groups by drawing one of two nontransparent envelopes which contained one ticket inscribed with either a E (for Euglyca group) or a C (for Control group). To ensure equal allocation rates within the 2 groups, block randomization was employed.

At the initial visit, patients randomized to the E group were advised to download the Euglyca application on their smartphones and they were asked to use the application for the calculation of the bolus insulin dose they were injected. Patients randomized to the C group were advised to calculate bolus insulin dose they were injected, the way they used to do. Patients repeated their visit to the endocrine pediatric clinic at 3, 6 and 12 months, the latter set as the terminal time-point of this study following the initial visit. At all 4 visits, anthropometrics (weight, height, BMI), blood pressure measurement and heart rate were noted down, while a peripheral blood sample was drawn from all patients in the morning of each visit after an overnight fast for measurement of glycemia and glycosylated hemoglobin (HbA1c) levels. Glucose measurements between 70 and 180 mg/dl were categorized as normoglycemia; any glucose measurement below 70mg/dl was categorized as hypoglycemia; glucose measurements at two hours postprandial measurement found above 180mg/dl were categorized as hyperglycemia. At baseline (first visit), at 6 months (third visit) and at terminal time-point (12 months) all patients filled the World Health Organization-Standard DTSQ. Patients' logbooks and readings from their glucose meters were reviewed by the physicians and nutritionist of the department at each of the four visits and the percentage of normoglycemic, hypoglycemic and hyperglycemic episodes during the preceding trimester was calculated for each patient. The change of HbA1c values from baseline to the terminal time-point for each group was set as primary outcome, while the percentage of normoglycemic, hypoglycemic and hyperglycemic events over the total number of glucose measurements during the preceding trimester of each visit was set as secondary outcome.

Glycosylated hemoglobin was determined by Siemens DCA Vantage point-of-care immunoassay analyzer (Siemens Health care Diagnostics Ltd., Frimley, Camberley, UK) with intra- and inter- assay coefficients of variation (CV) 5% and 8%, respectively; glycemia was determined by glucose god/pap kit with intra- and inter- assay CVs 5.7% and 7.8%, respectively.

'Euglyca' is a mobile application that we developed . The application has a data base of 7000 foods and food products met in greek eating habits as well as the corresponding amount of carbohydrates and lipids for each of them. Subsequently, the amount of carbohydrates and lipids contained in a meal are calculated automatically by the application. By taking into consideration the amount of carbohydrates and lipids to be consumed, the preprandial and target post-prandial glycemia concentrations, the insulin correction factor for the patient, the carbohydrates and lipids factors and the active insulin (in case of CSII), 'Euglyca' calculates the required bolus dose of insulin.

Sample size was determined by estimating the change in HbA1c values (primary outcome) based on previous studies (7, 8), assuming 0.5% reduction in HbA1c in the intervention group with 80% power and 5% significance level. Power calculation resulted in 14 patients per group, while the target of the study had been set at recruitment of 80 patients altogether. Results are reported as mean ± standard deviation (SD) for quantitative variables. The absolute difference in a quantitative variable between two different time points was defined as Δ. All quantitative variables (HbA1c; ΔHbA1c; percentages of normoglycemic, hypoglycemic and hyperglycemic events over a total number of glucose measurements; DTSQ's scores) were normally distributed and they were compared between the two studied groups of patients at the different time-points by employing General Linear Models ANOVA and Bonferroni post-hoc test. Repeated measures ANOVA involved one factor between patients (factor "Group" with two levels) and one factor for the repeated measures within patients (factor "time" with 4 or 3 levels depending on the compared variable). Qualitative variables (gender and type of therapy) were compared by employing x2 (chi square) test after having computed absolute and relative frequencies (percentages %), Statistical significance was set at P<0,05. An intention to treat analysis was followed. IBM SPSS V23 Chicago, USA software was used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with Diabetes Mellitus type 1.
* Treatment with multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII)
* Satisfactory knowledge of the concept of carbohydrates and lipids counting

Exclusion Criteria:

* Use of another medical application for diabetes in the previous 3 months;
* Lack of capacity of reading greek.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Level of glycosylated hemoglobin in the 2 groups | At 3 months after the baseline visit
  Comparison of the level of glycosylated hemoglobin between the 2 groups
Level of glycosylated hemoglobin in the 2 groups | At 6 months after the baseline visit
  Comparison of the level of glycosylated hemoglobin between the 2 groups
Level of glycosylated hemoglobin in the 2 groups | At 12 months after the baseline visit
  Comparison of the level of glycosylated hemoglobin between the 2 groups
Change from Baseline glycosylated hemoglobin at 3 months in the 2 groups | At 3 months after the baseline visit
  Comparison of the differences in the level of glycosylated hemoglobin between the 2 groups
Change from 3 months glycosylated hemoglobin at 6 months in the 2 groups | At 6 months after the baseline visit
  Comparison of the differences in the level of glycosylated hemoglobin between the 2 groups
Change from 6 months glycosylated hemoglobin at 12 months in the 2 groups | At 12 months after the baseline visit
  Comparison of the differences in the level of glycosylated hemoglobin between the 2 groups

SECONDARY OUTCOMES:
Percentage of Normoglycemias in the 2 groups | At 3 months after the baseline visit
  Comparison of the percentage of Normoglycemias between the 2 groups
Percentage of Normoglycemias in the 2 groups | At 6 months after the baseline visit
  Comparison of the percentage of Normoglycemias between the 2 groups
Percentage of Normoglycemias in the 2 groups | At 12 months after the baseline visit
  Comparison of the percentage of Normoglycemias between the 2 groups
Diabetes Treatment Satisfaction Questionnaire (DTSQ) score in the 2 groups | At 3 months after the baseline visit
  Comparison of the Diabetes Treatment Satisfaction Questionnaire (DTSQ) score between the 2 groups.
  DTSQ consists of 8 elements. Each element can be graded in a scale from 0 to 6. Two of the elements concern the perceived hypoglycemia or hyperglycemia. By adding the grades of each of the rest 6 elements the DTSQ score is calculated.
Diabetes Treatment Satisfaction Questionnaire (DTSQ) score in the 2 groups | At 6 months after the baseline visit
  Comparison of the Diabetes Treatment Satisfaction Questionnaire (DTSQ) score between the 2 groups.
  DTSQ consists of 8 elements. Each element can be graded in a scale from 0 to 6. Two of the elements concern the perceived hypoglycemia or hyperglycemia. By adding the grades of each of the rest 6 elements the DTSQ score is calculated.
Diabetes Treatment Satisfaction Questionnaire (DTSQ) score in the 2 groups | At 12 months after the baseline visit
  Comparison of the Diabetes Treatment Satisfaction Questionnaire (DTSQ) score between the 2 groups.
  DTSQ consists of 8 elements. Each element can be graded in a scale from 0 to 6. Two of the elements concern the perceived hypoglycemia or hyperglycemia. By adding the grades of each of the rest 6 elements the DTSQ score is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrine Unit of 3rd Department of Pediatrics of Aristotle University of Thessaloniki, Hippokration General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT03763474/Prot_SAP_001.pdf